CLINICAL TRIAL: NCT04369768
Title: Restoration of Permanent Molars Affected With Molar-incisor-hypomineralization (MIH) Among a Group of Egyptian Children Using Composite Restorations or Preformed Metal Crowns: Two-arm Randomized Controlled Trial (Part I)
Brief Title: Restoration of Permanent Molars Affected With Molar-incisor-hypomineralization (MIH) Among a Group of Egyptian Children Using Composite Restorations or Preformed Metal Crowns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sandra Nasr Fares, Dr. Sandra Nasr Fares, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIH restoration
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- direct composite restorations (Active Comparator)
  Interventions: Procedure: restoration of permanent molars affected with MIH
- preformed metal crowns (Active Comparator)
  Interventions: Procedure: restoration of permanent molars affected with MIH

INTERVENTIONS:
Procedure: restoration of permanent molars affected with MIH — restore MIH affected molars using direct composite or preformed metal crowns

SUMMARY:
The aim of this study is to compare the clinical outcome of using direct esthetic composite restorations and the use of preformed metal crowns in managing MIH cases among a group of Egyptian children.

ELIGIBILITY:
Inclusion Criteria:

* Children with MIH in one fully erupted molar or more.
* Age ranging from 7-12 years.
* Cooperative children
* Good general health.

Exclusion Criteria:

* patients participating in other experiments.
* Patients with parents planning to move away within the following year.
* Patients with only mildly affected MIH molars that do not require extensive restorative treatment.
* MIH-affected molars that have a very poor prognosis and require extraction.
* First permanent molars that are affected with other developmental defects, such as hypoplasia, dental fluorosis or amelogenesis imperfecta

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
treating hypersensitivity associated with MIH affected permanent molars by questioning the patient | one year
  questioning the patient about hypersensitivity after performing treatment ( direct composite restorations and preformed metal crowns)